CLINICAL TRIAL: NCT02543229
Title: A Phase 1 Dose Escalation Study Evaluating the Safety, Pharmacokinetics and Pharmacodynamics of OPT-302 in Combination With Ranibizumab in Subjects With Wet AMD
Brief Title: Study Evaluating the Safety, Pharmacokinetics and Pharmacodynamics of OPT-302 With or Without Lucentis™ in Patients With Wet AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Opthea Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPT-302-1001
Record Dates: First submitted 2015-08-25; First posted 2015-09-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Eye Diseases; Macular Degeneration; Retinal Diseases; Retinal Degeneration; Neovascularization, Pathologic
MeSH Terms: conditions — Eye Diseases; Macular Degeneration; Retinal Diseases; Retinal Degeneration; Neovascularization, Pathologic | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Part 1 Dose escalation - Cohort 1 (Experimental): Dose Level 1 of OPT-302 in combination with Lucentis™
  Interventions: Drug: OPT-302; Drug: Lucentis™
- Part 1 Dose escalation - Cohort 2 (Experimental): Dose Level 2 of OPT-302 in combination with Lucentis™
  Interventions: Drug: OPT-302; Drug: Lucentis™
- Part 1 Dose escalation - Cohort 3 (Experimental): Dose Level 3 of OPT-302 in combination with Lucentis™
  Interventions: Drug: OPT-302; Drug: Lucentis™
- Part 1 Dose escalation - Cohort 4 (Experimental): Dose Level 3 of OPT-302 monotherapy
  Interventions: Drug: OPT-302
- Part 2 Dose expansion - Cohort 5 (Experimental): OPT-302 (at Maximum Tolerated Dose [MTD] or highest dose tested in Part 1) in combination with Lucentis™
  Interventions: Drug: OPT-302; Drug: Lucentis™
- Part 2 Dose expansion - Cohort 6 (Experimental): OPT-302 (at MTD or highest dose tested in Part 1) monotherapy
  Interventions: Drug: OPT-302

INTERVENTIONS:
Drug: OPT-302 — OPT-302 will be administered by intravitreal injection once every month for 3 months
Drug: Lucentis™ — Lucentis™ (0.5 mg) will be administered by intravitreal injection once every month for 3 months
  Other Names: Ranibizumab
  Arms: Part 1 Dose escalation - Cohort 1; Part 1 Dose escalation - Cohort 2; Part 1 Dose escalation - Cohort 3; Part 2 Dose expansion - Cohort 5

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety, pharmacokinetics (PK) and pharmacodynamics of OPT-302 administered as monthly intravitreal injections for 3 months with and without Lucentis™ in patients with wet age related macular degeneration (AMD). This study will be conducted in two parts: Part 1 will comprise an open label, sequential dose escalation and Part 2 a randomized dose expansion.

OPT-302 is a soluble form of VEGFR-3 comprising the extracellular domains 1-3 of human vascular endothelial growth factor receptor (VEGFR)-3 and the Fc fragment of human IgG1. It functions by binding and neutralizing the activity of vascular endothelial growth factor (VEGF)-C and VEGF-D on endogenous VEGFR-2 and VEGFR-3.

VEGF-C and VEGF-D promote blood vessel development (angiogenesis) by binding and activating VEGFR-2 and VEGFR-3. VEGF-C is also a potent inducer of vascular permeability or leakage. Angiogenesis and vascular leakage are key hallmarks of wet AMD. Approved therapies for wet AMD include Eylea™ and Lucentis™ which block the activity of VEGF-A, but not VEGF-C or VEGF-D which are alternate members of the same family of molecules.

VEGF-C and VEGF-D can stimulate blood vessel growth and leakage through the same pathway as VEGF-A (via VEGFR-2), as well as through pathways that are independent of VEGF-A (via VEGFR-3). Published studies have also indicated that VEGF-C and VEGF-D play an important role in mediating resistance to therapies that block VEGF-A such as Lucentis™ and Eylea™.

Combination therapy with OPT-302 an anti-VEGF-A agent provides a more complete blockade of the VEGF family. This strategy targets functional redundancy in the VEGF pathway and mechanisms of 'resistance' or sub-response to VEGF-A inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Age ≥ 50 years of either gender
* Active CNV lesions secondary to AMD (i.e., subretinal or intraretinal fluid on SD-OCT and / or leakage on fluorescein angiography)
* Either no previous treatment in the study eye with IVT anti-VEGF-A therapy (treatment naïve) or prior IVT anti-VEGF-A therapy (previously treated) with sub-optimal response to treatment and the need for additional treatment
* Best corrected visual acuity in the study eye, using ETDRS testing, of 20/320 or better (Snellen equivalent) in Part 1 (dose escalation) and between 20/40 and 20/320 (Snellen equivalent), inclusive, in Part 2 (dose expansion).
* Women of child bearing potential and male subjects with female partners of child bearing potential must be practicing effective contraception during the trial and for at least 3 months following the last dose of study medication

Exclusion Criteria:

* Previous or concurrent use of systemic anti-VEGF-A agents
* Most recent IVT injection of bevacizumab or ranibizumab <28 days prior to screening or aflibercept <42 days prior to screening
* Previous treatment with photodynamic therapy, thermal laser or external beam radiation in the study eye
* Concurrent treatment in either eye for any ocular condition with an investigational drug or device that has not received regulatory approval
* Anatomic damage to the center of the fovea including fibrosis and scarring making up >50% of total lesion area including the CNV in the study eye
* Geographic atrophy involving the center of the fovea in the study eye
* History or presence of a retinal pigment epithelial tear
* Presence of polypoidal choroidal vasculopathy (if in the opinion of the investigator, anti-VEGF treatment would not be of benefit) or retinal angiomatous proliferation
* Active or recent (within 4 weeks) intraocular inflammation (grade trace or above) in the study eye
* History of rhegmatogenous retinal detachment or macular hole in the study eye
* History of vitrectomy
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* History of vitreous hemorrhage within 4 weeks prior to screening in the study eye
* History of major ocular surgery within prior 6 months or anticipated within next 3 months following dosing on day 1
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure of >25 mmHg despite treatment with maximal medical therapy)
* Uncontrolled hypertension ≥180 mmHg systolic or ≥110 mmHg diastolic at baseline
* Uncontrolled diabetes mellitus (Disease must be controlled with hemoglobin A1c (HgbA1c) < 9.0%)
* Clinical evidence of diabetic retinopathies, diabetic macular edema or any other vascular disease affecting the retina, other than AMD, in either eye that, in the opinion of the investigator, would be likely to limit improvement in the macular anatomy and/or function
* Pregnancy or lactation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-07; Primary Completion 2017-02-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse Events) | Up to 1 month after the last dose
  Subject incidences of ophthalmic and systemic Adverse Events during study and follow-up period

SECONDARY OUTCOMES:
Mean change in Best Corrected Visual Acuity (BCVA) from baseline | 6 months
  Mean change in Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA from baseline
Mean change in central retinal thickness from baseline | 6 months
  Changes in intra- or sub-retinal fluid measured as mean change in central retinal thickness or macula volume by Spectral Domain Optical Coherence Tomography (SD-OCT)
Mean change in Choroidal Neovascularization (CNV) lesion area from baseline | 6 months
  Change in CNV size according to fluorescein angiogram
Mean number of retreatment injections of anti-VEGF-A therapy during long term follow-up (week 12 to 24) | 3 months
Need for 'rescue therapy' with ranibizumab in subjects receiving OPT-302 monotherapy | 3 months
Assess the Pharmacokinetic profile of OPT-302 alone and in combination with ranibizumab following intravitreal administration | Up to 28 days post-dose
  Mean systemic OPT-302 Concentration-Time profile
Anti-OPT-302 antibody formation | Pre-dose and up to 3 months post-dose
  Incidence of anti-OPT-302 antibody formation

OTHER OUTCOMES:
Exploratory: Changes in the systemic blood levels of angiogenesis-related biomarkers | 3 months
  Change in systemic blood levels of angiogenesis-related biomarkers including, but not limited to: Vascular Endothelial Growth Factor A (VEGF-A), VEGF-C, VEGF-D, soluble VEGFR-2 and soluble VEGFR-3.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research, Study Director — Opthea Limited
Locations (14):
- United States (14):
  - Opthea Investigative Site, Phoenix, Arizona
  - Opthea Investigative Site, Beverly Hills, California
  - Opthea Investigative Site, Sacramento, California
  - Opthea Investigative Site, Santa Maria, California
  - Opthea Investigative Site, Fort Myers, Florida
  - Opthea Investigative Site, Pensacola, Florida
  - Opthea Investigative Site, Winter Haven, Florida
  - Opthea Investigative Site, Wichita, Kansas
  - Opthea Investigative Site, Bloomfield, New Jersey
  - Opthea Investigative Site, Charlotte, North Carolina
  - Opthea Investigative Site, Cleveland, Ohio
  - Opthea Investigative Site, West Columbia, South Carolina
  - Opthea Investigative Site, Abilene, Texas
  - Opthea Investigative Site, Willow Park, Texas